CLINICAL TRIAL: NCT02062515
Title: Safety Assessment of Icotinib in Advanced NSCLC Patients With Hepatic Insufficiency: A Multi-center, Open-label, Single-arm Study
Brief Title: Icotinib in Advanced Non-small Cell Lung Cancer (NSCLC) With Hepatic Insufficiency
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV51
Record Dates: First submitted 2014-02-12; First posted 2014-02-13 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Icotinib (Experimental): Icotinib is administered orally 125 mg three times per day continuously for four weeks
  Interventions: Drug: icotinib

INTERVENTIONS:
Drug: icotinib — Icotinib is administered orally 125 mg three times per day continuously for four weeks
  Other Names: BPI-2009; Commana

SUMMARY:
The purpose of this study is to determine whether Icotinib is efficient and safe in treating advanced non-small cell lung cancer (NSCLC) patients with hepatic insufficiency.

DETAILED DESCRIPTION:
Patients with hepatic insufficiency is an important subgroup of who receive EGFR TKIs. Phase I/II studies showed that Icotinib has good security. Based on the above considerations, this single-arm, open-label study is designed to evaluate the safety of icotinib 125mg three times daily for histologically or cytologically confirmed NSCLC patients with hepatic insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of IIIB/IV stage NSCLC patients who are not suitable for surgery or radiotherapy
* ECOG performance status points (PS) is 0-2
* Liver function:

A (mild hepatic dysfunction):

A1) total bilirubin within normal limit (ULN), while AST> ULN;

A2) total bilirubin within1.0-1 .5 × ULN;

B (moderate hepatic dysfunction): total bilirubin within1.5-3 .0 × ULN

* No malabsorption or other gastrointestinal disorders effecting drug absorption
* Life expectancy: more than 12 weeks.

Exclusion Criteria:

* Previous usage of HER/EGFR inhibitors or other target molecule drugs ( small molecule drugs or monoclonal antibody therapy )
* Patients requires liver shunt , stent placement, or radiotherapy when 2 weeks before the start of the study or research process .
* Patients with active hepatitis and cirrhosis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hao Long, MD, Principal Investigator — Sun Yat-sen Cancer Center
Locations (1):
- Sun Yat-sen Cancer Center, Guangzhou, Guangdong, China